CLINICAL TRIAL: NCT05681312
Title: Evaluation of the Effect of Systemic Proteolytic Enzyme Therapy on Postoperative Inflammatory Response and Quality of Life After Surgical Extraction of Impacted Mandibular Third Molars
Brief Title: Evaluation of the Effect of Systemic Proteolytic Enzyme Therapy on Postoperative Inflammatory Response and QoL After Surgical Extraction of Impacted Mandibular Third Molars
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Dunya Abdulmuniem, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 673122
Record Dates: First submitted 2022-12-13; First posted 2023-01-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain
Keywords: systemic proteolytic enzyme; pain; trismus; swelling; tibrolin
MeSH Terms: conditions — Pain, Postoperative; Pain; Trismus | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Tibrolin combination of (Trypsin 48 mg, Bromelain 90 mgand a bioflavonoid (Rutoside 100 mg) .one by one for five day
Who Masked: Participant
Masking Description: metronidazol 500 mg 1bythree amoxicillin 500 mg 1by three doulprane 1000 mg one by one
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemic proteolytic enzyme (Active Comparator): Tibrolin combination of (Trypsin 48 mg, Bromelain 90 mg) and a bioflavonoid (Rutoside 100 mg) one by one for five day
  Interventions: Drug: systemic proteolytic enzyme (Tibrolin)
- amoxicillin, metronidazol, doliprane (Placebo Comparator): amoxicillin 500 mg one by three metronidazol 500 mg one by three doulprane 1000 mg one by one
  Interventions: Drug: Amoxicillin 500mg+metronidazole 500mg+ doliprane 100mg

INTERVENTIONS:
Drug: systemic proteolytic enzyme (Tibrolin) — Tibrolin is a fixed dose combination of(Trypsin 48 mg, Bromelain 90 mg) and a bioflavonoid (Rutoside 100 mg)
  Other Names: tibrolin
  Arms: systemic proteolytic enzyme
Drug: Amoxicillin 500mg+metronidazole 500mg+ doliprane 100mg — Amoxicillin is given with metronidazole 500mg 1*3' Doliprane 1000mg is given 1*1
  Arms: amoxicillin, metronidazol, doliprane

SUMMARY:
1. To compare the postoperative pain between the patients who receive the systemic enzyme therapy and patients in the control group in the third and seventh day.
2. To compare the postoperative swelling (edema) between the patients who receive the systemic enzyme therapy and patients in the control group in the third and seventh day.
3. To compare the degree of trismus between the patients who receive the systemic enzyme therapy and patients in the control group in the third and seventh day.
4. Measure patients' perceptions of changes in their quality of life in the postoperative period and compare it between the patients who receive the systemic enzyme therapy and patients in the control group in the third and seventh day.

DETAILED DESCRIPTION:
Evaluation of the effect of systemic proteolytic enzyme therapy on postoperative inflammatory response and quality of life after surgical extraction of impacted mandibular third molar.

The aim of this study is to evaluate the effect of systemic enzyme therapy(TibrolinTM) on the postoperative inflammatory response and the quality of life after surgical removal of impacted third molar. The study is designed and was implemented as a randomized controlled clinical study guided by Consolidated Standards of Reporting Trials (CONSORT) guidelines . Patients were randomly allocated to two groups (25patients per group). Group A included administration of SET after surgery and continued for 5 days post-surgery; Group B, a control group that would not receive the systemic enzyme therapy . The predictor variable was The use of systemic proteolytic enzyme (Tibrolin) or not .The primary outcome variables were pain and swelling , trismus,quality of life measured on 1st day (day of surgery), third day, and 7th after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients over 18 years old of either gender.
* Patients who have impacted mandibular third molar.
* Ability to tolerate surgical procedure.
* Pell and Gregory's classification (Class I and class II, position A and B).

Exclusion Criteria:

* Patients with uncontrolled systemic diseases.
* Patients with history of chemotherapy or radiotherapy therapy to the head and neck region.
* Acute infection at the surgical site at time of operation.
* The presence of cysts or tumors associated with the impacted teeth.
* Pell and Gregory's classification (class III Position C)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-05-08 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Pain after surgery | 7 Days
  pain will be measured on pain rating scale form 0 to 10
Facial swelling | 7 Days
  swelling will be determined by distance between 3 points
Trismus | 7 Days
  the degree of trismus will be measured by maximum mouth opening

CONTACTS AND LOCATIONS:
Overall Officials: salwan bede, Study Director — University of Baghdad
Locations (1):
- Dunya Abdulmuniem Mahmood, Baghdad, Iraq